CLINICAL TRIAL: NCT03888560
Title: Duration Of Lower Labial Segment Alignment With Repeated Micro-Osteoperforations: Randomised Controlled Clinical Trial
Brief Title: Duration Of Lower Labial Segment Alignment With Repeated Micro-Osteoperforations:
Acronym: MOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGD170005
Record Dates: First submitted 2019-03-13; First posted 2019-03-25 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Malocclusion
Keywords: micro-osteperforation; orthodontic tooth movement; treatment duration
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: The start date of lower labial segment alignment (T1) was recorded after insertion of the lower 0.014'' NiTi archwire. Participants were reviewed every 6 weeks and repeated MOPs were performed for the MOP group until the completion of lower labial segment alignment (LLS), which is when the LII scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine. At the end of alignment stage, the date for completion of alignment was recorded (T2), from which the overall alignment time (OAT) in days, required to complete LLS alignment, were calculated. Measurements were done clinically using an electric digital caliper. At this point, perforations were stopped. Gingival recession and black triangle were then recorded and measured. Patients were referred for CBCT images to evaluate for root resorption.
Who Masked: Outcomes Assessor
Masking Description: Blinding of either patient or clinician is not possible during allocation, treatment and data collection. However, blinding can be ensured during data processing, analysing stages and data collection for secondary outcomes on total volume of root resorption from CBCT, formation of black triangle and gingiva recession
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-osteoperforations (Experimental): Lower arch, 2 MOPs vertically at interdental area bilaterally mesial to lower 6's ; mesial to lower 1st premolar; mesial to lower 2's and between the lower 1's..The start date of lower labial segment alignment (T1) was recorded after insertion of the lower 0.014'' NiTi archwire. Participants were reviewed every 6 weeks and repeated MOPs were performed for the experimental group until the completion of lower labial segment alignment (LLS), which is when the Little's irregularity index scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine.
  Interventions: Device: Micro-osteoperforations
- control (No Intervention): Conventional orthodontic treatment without any aid in tooth acceleration method / device

INTERVENTIONS:
Device: Micro-osteoperforations — MOPs will be performed using SIA Excalibur Mini-Implant with dimension 1.6 mm in width and length of 6 mm, screw 3 mm depth into buccal bone of intervention sites
  Arms: Micro-osteoperforations

SUMMARY:
The main purpose is to compare overall alignment time (OAT) in days in alleviating mandibular incisors crowding between control group and MOPs group.Furthermore, to investigate the presence of volumetric root resorption from CBCT, gingival recession and formation of black triangle post lower labial segment alignment between micro-osteoperforations group and control group.

DETAILED DESCRIPTION:
Prolonged treatment time in orthodontics is an undesirable side effect for both the patient and clinician. Usually, an average course of comprehensive orthodontic treatment with fixed appliances requires less than 2 years to complete (19.9 months). This prolonged treatment time may cause adverse effects such as root resorption, gingival recession, caries & enamel demineralization. Micro-osteoperforations is safe, minimally invasive technique which perforations are performed through the gum tissues, penetrating the bone without the need to raise a ﬂap.Control group will not received any MOP and will receive standard orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gender : Male and Female
* Age range : ≥ 18years to 45 years old
* Crowding of 3mm - 7mm on lower labial segment (lower right canine to lower left canine) which does not require extractions in the lower arch
* Class II div I Incisor relationship with extraction of both upper 1st premolars
* Maximum anchorage control with temporary anchorage device ( TAD) , with Molar Class II (¼ to full unit) malocclusion
* Average vertical facial proportions
* No systemic disease
* Acceptable good oral hygiene
* No periodontal disease

Exclusion Criteria:

* Smokers
* Distally angulated canines
* History of trauma (crown fracture or avulsion and re-implantation) , endodontic treatment
* Missing permanent mandibular anterior teeth ( Hypodontia) / Retained deciduous teeth in mandibular anterior area
* Habits eg: fingernails biting , toothpick user , using hard toothbrush
* Vertical skeletal discrepancies eg high angle and low angle
* Systemic disease especially on long term use of antibiotics, phenytoin, cyclosporin, anti-inflammatory drugs, systemic corticosteroid and calcium channel blockers
* Poor oral hygiene for more than 3 visits
* Current periodontal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
1. To compare the duration to align the lower labial segment (33-43), between regular and irregular review groups from the conventional (control group). | 5 months
  Total treatment time needed to achieved lower labial segment alignment until Little's irregularity index scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine
2. To compare the duration to align the lower labial segment (33-43), between regular and irregular review groups from the micro-osteoperforations group. | 5 months
  Total treatment time needed to achieved lower labial segment alignment until Little's irregularity index scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine
3. To compare the duration to align the lower labial segment (33-43), between micro-osteoperforations and control group in the regular review group. | 5 months
  Total treatment time needed to achieved lower labial segment alignment until Little's irregularity index scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine
4. To compare the duration to align the lower labial segment (33-43), between micro-osteoperforations and control group in the irregular review group. | 5 months
  Total treatment time needed to achieved lower labial segment alignment until Little's irregularity index scores one, indicating a minimum irregularity of ≤ 2 mm contact point displacement, based on the contact point displacements of the mandibular anterior segment, from canine to canine

SECONDARY OUTCOMES:
Total volume of root resorption with micro-osteoperforations group vs the control group | 5 months
  Total volume of root resorption in cubic millimeter (mm3) using 3D Cone Beam CT imaging scanner compare at baseline and end of LLS alignment
Gingival recession between micro-osteoperforations and control group. | 5 months
  Gingival recession assessed in millimetre (mm) from cement-enamel junction (CEJ) to free gingival margin using electric digital calliper with an accuracy of 0.01mm, at baseline and end LLS alignment
Black triangle between micro-osteoperforations and control group. | 5 months
  Presence of black triangle for interdental at baseline and end of LLS alignment

CONTACTS AND LOCATIONS:
Overall Officials: Nik Nuraini Nik Azmin, Principal Investigator — University of Malaya; lorretha p ringgingon, Principal Investigator — faculty of dentistry university of malaya; Saritha Sivarajan, Study Director — faculty of dentistry university of malaya; wey mang chek, Study Director — faculty of dentistry university of malaya; mona fayed, Study Director — faculty of dentistry university of malaya
Locations (1):
- Faculty of Dentistry , University of Malaya, Kajang, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixeira CC, Khoo E, Tran J, Chartres I, Liu Y, Thant LM, Khabensky I, Gart LP, Cisneros G, Alikhani M. Cytokine expression and accelerated tooth movement. J Dent Res. 2010 Oct;89(10):1135-41. doi: 10.1177/0022034510373764. Epub 2010 Jul 16. PMID 20639508
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] Alkebsi A, Al-Maaitah E, Al-Shorman H, Abu Alhaija E. Three-dimensional assessment of the effect of micro-osteoperforations on the rate of tooth movement during canine retraction in adults with Class II malocclusion: A randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):771-785. doi: 10.1016/j.ajodo.2017.11.026. PMID 29853235
- [Background] Sivarajan S, Doss JG, Papageorgiou SN, Cobourne MT, Wey MC. Mini-implant supported canine retraction with micro-osteoperforation: A split-mouth randomized clinical trial. Angle Orthod. 2019 Mar;89(2):183-189. doi: 10.2319/011518-47.1. Epub 2018 Oct 29. PMID 30372126
- [Background] Attri S, Mittal R, Batra P, Sonar S, Sharma K, Raghavan S, Rai KS. Comparison of rate of tooth movement and pain perception during accelerated tooth movement associated with conventional fixed appliances with micro-osteoperforations - a randomised controlled trial. J Orthod. 2018 Dec;45(4):225-233. doi: 10.1080/14653125.2018.1528746. Epub 2018 Oct 3. PMID 30281397